CLINICAL TRIAL: NCT05347290
Title: Comparison Of Effective Radiation Shielding Between A Portable, Configurable, Floor-Supported Radiation Protection System vs Conventional Apron And Shields In Clinical Interventional Procedures
Brief Title: Comparison Of Effective Radiation Shielding Between Rampart IC, M1128 Shield vs Conventional Apron And Shields In Clinical Interventional Procedures
Acronym: RAMPART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Varinder Singh, Senior Vice President, Cardiology, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-1302
Record Dates: First submitted 2022-03-31; First posted 2022-04-26 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Radiation Exposure
Keywords: radiation; radiation exposure; interventional cardiology; cardiac catherization laboratory; cardiac cath lab; lead apron; RAMPART Shield; radiation protection

STUDY DESIGN:
Intervention Model Description: This single center randomized 1-3 month clinical study compares conventional lead aprons and ancillary shields to the Rampart IC, M1128 fully configurable, portable, floor supported system that provides radiation protection and orthopedic safety for operators and the scrubbed interventional team members. There will be three study arms, each arm requiring 21 procedures for a total of 63 total procedures. Each enrolled subject may be involved in more than one procedure/case. For all arms, subjects will wear real-time dosimeters on their right temple, shoulder, and hip, and values will be collected post-procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Lead Apron + Rampart IC, M1128 (Experimental): Consented providers will perform catherization procedures utilizing both lead apron and Rampart system. Radiation will be measured by dosimeters worn by the providers.
  Interventions: Device: Rampart IC, M1128 and Lead Apron
- Rampart M1128 IC, Only (Experimental): Consented providers will perform catherization procedures utilizing only the Rampart system. Radiation will be measured by dosimeters worn by the providers.
  Interventions: Device: Rampart IC, M1128
- Lead Apron Only (Active Comparator): This is the control group. Consented providers will perform catherization procedures utilizing only the lead apron and ancillary shields (lead skirt, vest, thyroid collar (all at least 0.5mm Pb) with use of under table lead per lab operating policy and mobile suspended lead-acrylic shield and lead glasses). Radiation will be measured by dosimeters worn by the providers.
  Interventions: Device: Lead Apron and Ancillary Shield

INTERVENTIONS:
Device: Rampart IC, M1128 — Rampart IC, M1128 aims to address the challenge of radiation protection in the cardiac catheterization laboratory without the burden of wearing a heavy lead apron. Rampart M1128 is a compactly designed, portable, fully adjustable system that provides radiation protection for interventionalists and their technicians. It has independently adjustable flexible panels, allowing interventionalists multiple vascular access points, including right radial, bi-lateral femoral, and bi-lateral pedal. Participants in this arm will conduct catherization procedures using only the Rampart System, and radiation exposure will be measured using real-time dosimeters.
  Other Names: Rampart Shield; Rampart; Rampart System; Rampart M1128
  Arms: Rampart M1128 IC, Only
Device: Lead Apron and Ancillary Shield — Participating providers in this arm will use conventional skirt and vest, thyroid collar, and 100% use of 2 types of ancillary shields. Most wrap-around skirts and vests were (0.25-0.5 mm) Pb. Thyroid shields were 0.5 mm Pb equivalent. Under the table lead x 2. Radiation exposure will be measured using real-time dosimeters.
  Other Names: LAS; Lead Apron
  Arms: Lead Apron Only
Device: Rampart IC, M1128 and Lead Apron — Participating providers will use both the lead apron and the Rampart Shield. Radiation exposure will be measured using real-time dosimeters.
  Arms: Lead Apron + Rampart IC, M1128

SUMMARY:
Previous studies have documented that orthopedic injuries and musculoskeletal pain are a likely result of wearing heavy leaded aprons. This single-center, randomized 1-3 month clinical study compares conventional lead aprons and ancillary shields to the Rampart IC, M1128 radiation protection system in order to improve radiation safety with minimal orthopedic strain by using the RAMPART device. There will be three study arms, each arm requiring 21 procedures for a total of 63 total procedures, Each procedure will be randomized, instead of individual subjects. Each enrolled subject may be involved in more than one procedure/case. Randomization stratification will be 1:1:1 to either Rampart shield only, lead apron and ancillary shield, or lead apron and Rampart Shield. Real-time dosimeters will be used in each procedure to measure radiation attenuation.

DETAILED DESCRIPTION:
Previous studies have documented that orthopedic injuries and musculoskeletal pain are a likely result of wearing heavy leaded aprons that are designed to shield interventionalists and laboratory staff from radiation. A large, multicenter study found that interventional laboratory employees reported a 67% increase in the prevalence of musculoskeletal pain. Two Society of Cardiovascular Angiography and Intervention (SCAI) surveys were performed a decade apart in 2004 and 2014 which both showed similar results on the orthopedic complications on the operators who wear leaded apron protection. The surveys revealed a 60% incidence of orthopedic issues and operators who have been operating greater than 20 years in the Cath Lab compared to a 2.3% incidence of chronic spine problems in the general population. Interestingly, of the operators who had been in practice less than 5 years, 26% already had orthopedic complaints. The study also revealed that over a third of those surveyed had already had to take spine related periods of absence from the catheterization lab. Though in recent years focus on individual radiation attenuation technologies that support both attenuation and orthopedic safety have evolved, the emphasis has been on the operator. A solution has not existed to address radiation attenuation and orthopedic safety for the entire scrubbed interventional team with one system.

To address the challenge of radiation protection in this environment without the burden of wearing a heavy lead apron, Rampart IC, M1128 was created. Rampart IC, M1128 is a fully adjustable and portable system that provides radiation protection for operators and their team without having to wear a lead apron. This study will have three randomization arms, each arm requiring 21 procedures for a total of 63 total procedures. Randomization stratification will be based on procedure, not individual subject. Each enrolled subject may be involved in more than one procedure/case. Computer software will be utilized to randomize procedures in a 1:1:1 ratio to either lead apron with ancillary shield, Rampart IC, M1128, or lead apron with the Rampart IC, M1128. Real-time dosimeters will be placed on interventional staff's left temple, shoulder, and hip in order to measure radiation attenuation.

ELIGIBILITY:
Inclusion Criteria:

* Participants > 18 years of age.
* Interventional cardiology staff at Lenox Hill Hospital that are scheduled to work in Room C of the cardiac catheterization laboratory.

Exclusion Criteria:

* Pregnancy
* Unwilling to consent to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Change in radiation attenuation | 90 days
  Change in radiation attenuation as detected by dosimeter readings for staff assigned to each randomization stratification.

CONTACTS AND LOCATIONS:
Overall Officials: Varinder P Singh, M.D., Principal Investigator — Senior Vice President, Cardiology
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Andreassi MG, Piccaluga E, Guagliumi G, Del Greco M, Gaita F, Picano E. Occupational Health Risks in Cardiac Catheterization Laboratory Workers. Circ Cardiovasc Interv. 2016 Apr;9(4):e003273. doi: 10.1161/CIRCINTERVENTIONS.115.003273. PMID 27072525
- [Background] Zakeri F, Hirobe T, Akbari Noghabi K. Biological effects of low-dose ionizing radiation exposure on interventional cardiologists. Occup Med (Lond). 2010 Sep;60(6):464-9. doi: 10.1093/occmed/kqq062. Epub 2010 Jun 2. PMID 20519631
- [Background] Klein LW, Miller DL, Balter S, Laskey W, Haines D, Norbash A, Mauro MA, Goldstein JA. Occupational health hazards in the interventional laboratory: time for a safer environment. Radiology. 2009 Feb;250(2):538-44. doi: 10.1148/radiol.2502082558. PMID 19188321
- [Background] Picano E, Vano E. The radiation issue in cardiology: the time for action is now. Cardiovasc Ultrasound. 2011 Nov 21;9:35. doi: 10.1186/1476-7120-9-35. PMID 22104562
- [Background] Orme NM, Rihal CS, Gulati R, Holmes DR Jr, Lennon RJ, Lewis BR, McPhail IR, Thielen KR, Pislaru SV, Sandhu GS, Singh M. Occupational health hazards of working in the interventional laboratory: a multisite case control study of physicians and allied staff. J Am Coll Cardiol. 2015 Mar 3;65(8):820-826. doi: 10.1016/j.jacc.2014.11.056. PMID 25720626
- [Background] Goldstein JA, Balter S, Cowley M, Hodgson J, Klein LW; Interventional Committee of the Society of Cardiovascular Interventions. Occupational hazards of interventional cardiologists: prevalence of orthopedic health problems in contemporary practice. Catheter Cardiovasc Interv. 2004 Dec;63(4):407-11. doi: 10.1002/ccd.20201. PMID 15558765
- [Background] Klein LW, Tra Y, Garratt KN, Powell W, Lopez-Cruz G, Chambers C, Goldstein JA; Society for Cardiovascular Angiography and Interventions. Occupational health hazards of interventional cardiologists in the current decade: Results of the 2014 SCAI membership survey. Catheter Cardiovasc Interv. 2015 Nov;86(5):913-24. doi: 10.1002/ccd.25927. Epub 2015 Mar 24. PMID 25810341
- [Background] Hirshfeld JW Jr, Balter S, Brinker JA, Kern MJ, Klein LW, Lindsay BD, Tommaso CL, Tracy CM, Wagner LK, Creager MA, Elnicki M, Lorell BH, Rodgers GP, Weitz HH; American College of Cardiology Foundation; American Heart Association/; HRS; SCAI; American College of Physicians Task Force on Clinical Competence and Training. ACCF/AHA/HRS/SCAI clinical competence statement on physician knowledge to optimize patient safety and image quality in fluoroscopically guided invasive cardiovascular procedures: a report of the American College of Cardiology Foundation/American Heart Association/American College of Physicians Task Force on Clinical Competence and Training. Circulation. 2005 Feb 1;111(4):511-32. doi: 10.1161/01.CIR.0000157946.29224.5D. No abstract available. PMID 15687141
- [Background] Ross AM, Segal J, Borenstein D, Jenkins E, Cho S. Prevalence of spinal disc disease among interventional cardiologists. Am J Cardiol. 1997 Jan 1;79(1):68-70. doi: 10.1016/s0002-9149(96)00678-9. PMID 9024739
- See also: Rampart IC, M1128 website — https://www.rampartic.com/